CLINICAL TRIAL: NCT05608447
Title: Effect and Safety of Intensive Fecal Microbiota Transplantation on Primary Hypertension: a Randomized Clinical Trial.
Brief Title: Effect of Intensive FMT on Primary Hypertension
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, Professor, Doctoral supervisor, Assistant Principal of Fuwai Hospital, Chief of Hypertension Center, Fuwai Hospital,PUMC&CAMS, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-GZ10 (Part III)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hypertension
Keywords: hypertension; microbiome; fecal microbiota transplantation; treatment
MeSH Terms: conditions — Hypertension | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT capsules (Active Comparator): FMT capsules containing extensively screened donor stool. FMT capsules will be orally taken on Day 0 (randomization), Day 1, Day 2, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49.
  Interventions: Biological: FMT capsules
- Placebo capsules (Placebo Comparator): Placebo capsules that do not contain donor stool or any active drug. Placebo capsules will be orally taken on Day 0 (randomization), Day 1, Day 2, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49.
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Biological: FMT capsules — FMT capsules containing extensively screened donor stool.
  Arms: FMT capsules
Other: Placebo capsules — Placebo capsules that do not contain donor stool or any active drug.
  Arms: Placebo capsules

SUMMARY:
Mounting preclinical and clinical evidences have proved the causal role of gut microbiota on the pathogenesis of primary hypertension. Restoration of gut microbiota ameliorated high BP in rodents and/or human cases.A hypothesis is thus raised that gut microbiome restoration can be a potential approach to ameliorate hypertension. This study will perform intense fecal microbiota transplantation (FMT) intervention via oral capsules, in comparison with placebo capsules, to investigate the effect, safety and underlying mechanisms of gut microbiome intervention on primary hypertension.

DETAILED DESCRIPTION:
Primary hypertension is a most prevalent cardiovascular diseases, and becomes a severe global public health issue because of the high morbidity and potential risk to other cardiovascular diseases. Several animal studies and diverse patient cohorts reported that the disorder of gut microbiome correlated with hypertension. Based on the investigators' previous work findings, a casual role of gut microbiome disorder was observed in primary hypertension (Microbiome. 2017;5(1):14.), and trend of ameliorating SBP was observed after short-course FMT intervention but recovery after intervention termination(Trials. 2022;23(1):178, unpublished results). The investigators therefore developed a consecutive study of intensive FMT intervention on primary hypertension.

Objective: To explore the effect, safety and underlying mechanisms of intensive FMT on primary hypertension.

Study Design: A multi-center, randomized, blinded, placebo-controlled pilot study.

Data quality control and statistical analysis: The investigators have invited professional statistic analysts to assist analyzing data and a third party to supervise data quality.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~65 years.
2. Established Diagnosis of Grade 1 Hypertension (initial diagnosis or free from antihypertensive drugs within a month): 140mmHg≤ Office SBP<160mmHg and/or 90mmHg≤ Office DBP<100mmHg for three measurements at different days without any antihypertensive medications, according to the"2010 Chinese Guidelines for Prevention and Treatment of Hypertension".
3. Patients with informed consent after thorough explanation.

Exclusion Criteria:

1. Antibiotics or probiotics usage within last 4 weeks
2. Participants of other clinical trials related to hypertension currently or within last 3 months
3. Antihypertensive medications usage currently or within last month
4. Diagnosed secondary hypertension
5. Severe hepatic or renal diseases ((ALT >3 times the upper limit of normal value, or end stage renal disease on dialysis or eGFR <30 mL/min/1.73 m2, or serum creatinine >2.5 mg/dl [>221 μmol/L])
6. History of large atherosclerotic cerebral infarction or hemorrhagic stroke(not including lacunar infarction and transient ischemic attack [TIA])
7. Hospitalization for myocardial infarction within last 6 months; Coronary revascularization (PCI or CABG) within last 12 months; Planned for PCI or CABG in the next 12 months.
8. Sustained atrial fibrillation or arrhythmias at recruitment disturbing the electronic BP measurement.
9. NYHA class III-IV heart failure; Hospitalization for chronic heart failure exacerbation within last 6 months.
10. Severe valvular diseases; Potential for surgery or percutaneous valve replacement within the study period.
11. Dilated cardiomyopathy; Hypertrophic cardiomyopathy; Rheumatic heart disease; Congenital heart disease.
12. Other severe diseases influencing the entry or survival of participants, such as malignant tumor or acquired immune deficiency syndrome.
13. Cognitive impairment or severe neuropsychiatric comorbidities who are incapable of providing their own informed consent.
14. Participants preparing for or under pregnancy and/or lactation.
15. Other conditions inappropriate for recruitment according to the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Office Systolic Blood Pressure (SBP) | From baseline to Week 8
  Change in Office Systolic Blood Pressure (SBP)

SECONDARY OUTCOMES:
Change in Office Systolic Blood Pressure (SBP) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 12
  Change in Office Systolic Blood Pressure (SBP)
Change in Office Diastolic Blood Pressure (DBP) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12
  Change in Office Diastolic Blood Pressure (DBP)
Change in Home Systolic Blood Pressure (SBP) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12
  Change in Home Systolic Blood Pressure (SBP)
Change in Home Diastolic Blood Pressure (DBP) | Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 12
  Change in Home Diastolic Blood Pressure (DBP), compared with baseline
Change in average SBP via 24-hour Ambulatory BP Monitoring | Baseline, Week 4, Week 8, Week 12
  Change in average SBP via 24-hour Ambulatory BP Monitoring
Change in average DBP via 24-hour Ambulatory BP Monitoring | Baseline, Week 4, Week 8, Week 12
  Change in average DBP via 24-hour Ambulatory BP Monitoring
Change in daytime SBP via 24-hour Ambulatory BP Monitoring | Baseline, Week 4, Week 8, Week 12
  Change in daytime SBP via 24-hour Ambulatory BP Monitoring
Change in daytime DBP via 24-hour Ambulatory BP Monitoring | Baseline, Week 4, Week 8, Week 12
  Change in daytime DBP via 24-hour Ambulatory BP Monitoring
Change in nighttime SBP via 24-hour Ambulatory BP Monitoring | Baseline, Week 4, Week 8, Week 12
  Change in nighttime SBP via 24-hour Ambulatory BP Monitoring
Change in nighttime DBP via 24-hour Ambulatory BP Monitoring | Baseline, Week 4, Week 8, Week 12
  Change in nighttime DBP via 24-hour Ambulatory BP Monitoring
Number of Participants with Adverse Events (AEs) as a Measure of Safety | All AEs over 12 weeks
  Number of Participants with Adverse Events (AEs) as a Measure of Safety
Changes in Intestinal Microbiota Composition Pre- and Post-intervention via Metagenomic Analysis | Baseline, Week 4, Week 8, Week 12
  Changes in Intestinal Microbiota Composition Pre- and Post-intervention (FMT or Placebo) via Metagenomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Changes in Intestinal Microbiota function revealed by KEGG pathways and KEGG Orthology (KO) Pre- and Post-intervention via Metagenomic Analysis | Baseline, Week 4, Week 8, Week 12
  Changes in Intestinal Microbiota function revealed by KEGG pathways and KEGG Orthology (KO) Pre- and Post-intervention via Metagenomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Durability of Engraftment of Donor Microbiome Following FMT | Baseline, Week 4, Week 8, Week 12
  Durability of engraftment of donor microbiome following FMT, measured by similarity comparison of intestinal microbiota composition between donor and recipient
Changes in Plasma Metabolite Composition Pre- and Post-intervention via Metabolomic Analysis | Baseline, Week 4, Week 8, Week 12
  Changes in Plasma Metabolite Composition Pre- and Post-intervention (FMT or Placebo) via Metabolomic Analysis, stratified by:
  1. Randomisation
  2. Change in Office SBP
Change in Fasting Blood Glucose Level | Baseline, Week 4, Week 8, Week 12
  Change in Fasting Blood Glucose Level
Change in blood HbA1c level | Baseline, Week 4, Week 8, Week 12
  Change in blood glycosylated hemoglobin, type A1C (HbA1c) level
Change in blood lipid level | Baseline, Week 4, Week 8, Week 12
  Change in Blood Lipid Level (Total Cholesterol, Total Triglyceride, Low Density Lipoprotein Cholesterol, High Density Lipoprotein Cholesterol)
Change in Body Mass Index | Baseline, Week 4, Week 8, Week 12
  Change in Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (3):
- China (3):
  - The Second Affiliated Hospital of Shantou University, Shantou, Guangdong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The People's Hospital of Ji Xian District, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
The collected data, study protocol, and SAP are planned to be shared after the study ends 2 years later (anticipated)
Supporting Information: Study Protocol, SAP
Time Frame: after the study ends 2 years later (anticipated)
Access Criteria: Access to these de-identified data will be required for written permission from the responsible investigation center and only for qualified researchers.

REFERENCES:
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Result] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Result] Fan L, Ren J, Chen Y, Wang Y, Guo Z, Bu P, Yang J, Ma W, Zhu B, Zhao Y, Cai J. Effect of fecal microbiota transplantation on primary hypertension and the underlying mechanism of gut microbiome restoration: protocol of a randomized, blinded, placebo-controlled study. Trials. 2022 Feb 24;23(1):178. doi: 10.1186/s13063-022-06086-2. PMID 35209934